CLINICAL TRIAL: NCT06673108
Title: Vaginal Photobiomodulation for Chronic Pelvic Pain: a Randomized Controlled Trial
Brief Title: Vaginal Photobiomodulation for Chronic Pelvic Pain
Acronym: VOICE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SoLa Pelvic Therapy (Industry)
Collaborators: Uroshape LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SoLaPelvicTherapy
Record Dates: First submitted 2024-10-25; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pelvic Pain; Chronic Pelvic Pain Syndrome (CPPS)
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Vaginal photobiomodulation (Active Comparator): Vaginal photobiomodulation with near-infrared (810-980nm wavelength) energy.
  Interventions: Device: SoLa Pelvic Therapy
- Sham-Light without laser energy. (Sham Comparator): Vaginal light therapy without focused laser energy.
  Interventions: Device: SoLa Pelvic Therapy

INTERVENTIONS:
Device: SoLa Pelvic Therapy — SoLa Pelvic Therapy laser emits near-infrared (810-980 nm wavelength) energy to the vaginal tissues. The device treats at 5-8 W for 3-6 minutes and delivers a fluence of 3,000 and 5,000 J/cm2 through a sterile vaginal probe. Specific treatment time is calculated based on vaginal length. Based on a code input, the device can cycle between emitting laser energy or sham which is visible light without focused laser energy.
  Other Names: Low level laser therapy

SUMMARY:
The goal of this clinical study is to determine if 8 treatments with photobiomodulation using near-infrared laser energy can help reduce chronic pelvic pain in women. Additionally, researchers want to determine if treatment with this type of energy can also alleviate pain with activities such as standing, sitting, urinating, having bowel movements and intercourse.

DETAILED DESCRIPTION:
This clinical trial will be a multi-center, triple-masked randomized study comparing vaginal photobiomodulation to sham, for the treatment of chronic pelvic pain in women. The study will include 126 participants, 63 randomized to vaginal photobiomodulation and 63 randomized to vaginal sham treatment. Potential participants will be recruited in communities and clinics where gynecologists are routinely evaluating patients for chronic pelvic pain.

Women who fulfill inclusion criteria will undergo, screening gynecologic evaluation to ensure they can participate. Informed and written consent will be obtained from all study participants prior to enrollment.

After consent, participants will be randomized to 8 treatments with active photobiomodulation or sham administered twice a week. Study subjects will be randomized using blocked 1:1 randomization with random permuted blocks of 4. Participants, study investigators, staff, and statisticians will remain masked throughout the study and unaware of whether sham or active laser is being administered to each participant.

Treatments will be administered using the SoLá Pelvic Therapy laser, which has been modified to emit sham or active photobiomodulation through the vagina using a thin laser wand protected by a sterile plastic covering. Treatments will be administered by a gynecology providers who specialize in evaluation and management of chronic pelvic pain. The SoLá Pelvic Therapy device auto-calculates power and duration of treatment based on vaginal length. The procedure typically lasts 3-6 minutes depending on the vaginal length and the pre-determined dosing selected by the device.

Patient reported pain levels will be assessed prior to each treatment and again at 1-week and 3-months after treatment. Pain levels will be obtained from both groups at baseline and after each treatment, while demographics, pain intensity, pain impact, pain behavior, and quality of life measures (QoL) will be collected at baseline and after treatment. Need for additional therapies, global impression of change, adherence and satisfaction will be assessed after 8 treatments. To assess effect duration, both groups will be followed for an additional 3 months, after which pain levels, QoL, use of additional treatments, global health, global impression of change, and satisfaction with the procedure will be assessed. After the 3-month follow-up, participation will come to an end.

The primary outcome will be to determine the percentage of participants who achieve a minimal clinically important difference (MCID) in overall pelvic pain, defined as a post-treatment decrease of ≥2 points on a 0-10 pain NRS (Numeric Rating Scale) at 3 months compared to baseline. Secondary outcomes include changes from baseline in:

* mean NRS pain levels of overall pelvic pain and symptom specific pelvic pain (pain with exercise, sitting, standing, bowel movements, urination, and intercourse);
* percentage of patients achieving MICD for symptom specific pelvic pain
* quality of life measured by decrease in pain intensity, impact, and interference, reduced need for additional treatments;
* improvement in global health;
* global impression of change,
* adherence and satisfaction with treatment. The intervention will be considered superior if 30% or higher percentage of participants achieve MCID compared to placebo (e.g., 30% in sham group vs 60%), or the intervention results in ≥1.1 NRS points reduction in mean pain levels compared to sham (e.g., intervention reduces mean pain levels by 2.4 points while sham reduces mean pain levels by 1.2 NRS points).

All patient reported outcomes (PROs) will be recorded using electronic surveys; many are specifically validated to measure pelvic pain, pelvic function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. CPP for 3 months or longer;
3. Overall pelvic pain severity ≥4 in the last 7 days;
4. Pelvic muscle tenderness pain level ≥4.

Exclusion Criteria:

1. Previous vaginal or vulvar laser therapy;
2. Receiving concurrent pelvic physical therapy;
3. Unable to tolerate vaginal/pelvic examination
4. Taking drugs that have heat- or light- sensitive contraindications;
5. Subjectively reports abnormal or decreased sensation in the vagina or rectum;
6. History of cancer of the cervix, vagina, uterus, bladder, or vulva or suspected of having neoplasia or pre-cancerous lesions;
7. History of autoimmune inflammatory conditions such as vulvar lichen sclerosis or other types of dermatoses;
8. History of vaginal trauma, ulcerations, erosions, or other evidence of vaginal and vulvar skin breakdown;
9. Less than 6 months post-partum;
10. Actively trying to get pregnant or not willing to use contraception during the trial;
11. Positive pregnancy test or planning to get pregnant during the study;
12. Vaginal discharge or bleeding concerning for neoplasia, infectious, or autoimmune condition; *
13. Pelvic pain has not been fully evaluated or pain is not confirmed as chronic pelvic pain;
14. Does not speak, read, or writes English and thus cannot complete surveys;
15. Does not have access to smart digital devices or computer, or cannot receive emails.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall pelvic pain | At baseline, at 1-week after completing treatment, and at 3 months after completing treatment.
  Overall pelvic pain level as measured on a 0-10 numeric rating pain scale (NRPS). On this scale, 0 represents no pain and 10 represents wors pain possible. Pain will be analyzed as median pain levels and % of participants achieving a minimal clinically important difference (MCID) defined as reduction in pain level of 2 or more NRPS points.

SECONDARY OUTCOMES:
Symptom specific pelvic pain | At baseline, at 1-week after completing treatment, and at 3 months after completing treatment.
  Pain with exercise, sitting, standing, bowel movements, urination, and intercourse as measured on a 0-10 numeric rating pain scale and analyzed in the same manner as the primary outcome 'overall pelvic pain'.
Pain impact | At baseline, at 1-week after completing treatment, and at 3 months after completing treatment.
  Pain intensity as measured by Patient Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Scale and Pain Interference Scale. The scales assess the impact of pain on activity, mood, relationships, sleep, and general enjoyment of life. The PROMIS Pain Intensity Scale asks participants to categorize pain intensity in the last 7 days, as an ordinal categorical scale using words like 'had no pain', 'mild', 'moderate', 'severe', and 'very severe', and the PROMIS Pain Interference Scale asks participants about the degree that pain interferes with activity, work around the home, participation in social activities, things usually done for fun, enjoyment of life, family life. Participants can rank their answers as an ordinal scale using words like 'not at all', 'a little bit', 'somewhat', 'quite a bit', and 'very much'.
Quality of life | At baseline, at 1-week after completing treatment, and at 3 months after completing treatment.
  As measured by the Short Form-12 Health Survey (SF-12), a self-reported outcome measure assessing the impact of health on an individual's everyday life. The SF-12 assess general health and well-being [or health-related quality of life (HRQOL)], including the impact of any and all illnesses on a broad range of functional domains. The SF-12 has two components scored on a range of 0-100: a physical component score (PCS) and a mental component score (MCS). A score of 50 or less on the PCS-12 indicates poor physical functioning or a physical condition, because scores above 50 indicate better than average health related quality of life, while a score below 50 suggests below average health. A score of 42 or less on the MCS-12 may indicate clinical depression. Therefore, SF-12 scores above 50 indicate better health and scores below 50 indicate worse than average health.
Global physical and mental health | At baseline, at 1-week after completing treatment, and at 3 months after completing treatment.
  Global physical and mental health as measured by the PROMIS Global Health questionnaire. It contains questions that allows participants to rank their general physical health, ability to carry out every day physical activities such as walking, climbing stairs, carry groceries, or moving a chair, using an ordinal scale ranking 'excellent', 'very good', 'good', 'fair', and 'poor'. This questionnaire also contains questions that allows participants to rate their mental health including ability to think, and satisfaction with social activities and relationships on an ordinal scale ranking 'excellent', 'very good', 'good', 'fair', and 'poor'.
Satisfaction with treatment. | At 1-week after completing treatment.
  Likert scale to describe satisfaction and likelihood of recommending treatment to a friend with a similar condition. Satisfaction is assessed with one question where participants are asked to rank their satisfaction with SoLa Pelvic Therapy on a Likert ordinal scale ranking satisfaction as 'very satisfied', 'satisfied', 'not satisfied', and 'very satisfied'. Likelihood of recommending the therapy to a friend is assessed with a Likert ordinal scale ranking 'very likely', 'somewhat likely', 'not likely', and 'very unlikely'.
Adherence with treatment. | After 5 treatments are completed.
  Measured as the percentage of completed treatments per participant and percentage of participants who completed 5 or more treatments.
Need for additional treatment | This questionnaire is completed once a week, prior to each treatment through administration of all 8 treatments (which are administered twice a week), and again at 3 months after completing the last treatment.
  Questionnaire that collects data on additional pharmacologic or non-pharmacologic, extra-pelvic, pain therapies used during the study duration (excluding laser and physical therapy).
Global impression of change | At 1-week after completing treatment, and at 3 months after completing treatment.
  a single, self-administered question asking respondents to rate whether their condition has changed after treatment compared to baseline before treatment. They are asked to select a response based on the following categories: 'very much improved', 'much improved', 'minimally improved', 'no change', 'minimally worse', 'much worse', and 'very much worse'.

CONTACTS AND LOCATIONS:
Overall Officials: Georgine Lamvu, MD, MPH, Principal Investigator — SoLá Pelvic Therapy
Locations (5):
- United States (5):
  - Obgyn South, Birmingham, Alabama
  - The Orady Womens Clinic, San Francisco, California
  - Urogynecology of Kansas City, Overland Park, Kansas
  - Boston Urogyn, Boston, Massachusetts
  - Nurture Women's Health, Frisco, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data tables may be shared after permission is obtained from the study sponsor.
Supporting Information: Study Protocol, ICF
Time Frame: After analysis and publication is complete and up to a period of 2 years.
Access Criteria: The study protocol and database will be available after express consent from the study sponsor.
URL: https://www.voiceclinicaltrial.com/

REFERENCES:
- [Background] Zipper R, Pryor B, Lamvu G. Transvaginal Photobiomodulation for the Treatment of Chronic Pelvic Pain: A Pilot Study. Womens Health Rep (New Rochelle). 2021 Nov 23;2(1):518-527. doi: 10.1089/whr.2021.0097. eCollection 2021. PMID 34841398
- [Background] Zipper R, Pryor B. Evaluation of a novel deep tissue transvaginal near-infrared laser and applicator in an ovine model. Lasers Med Sci. 2022 Feb;37(1):639-643. doi: 10.1007/s10103-021-03315-z. Epub 2021 Apr 14. PMID 33855615